CLINICAL TRIAL: NCT05341687
Title: Prognostic Value of Respiratory System Compliance Under VV-ECMO on 180-day Mortality in Patients With COVID-19 Associated Acute Respiratory Distress Syndrome (CARDS)
Brief Title: Prognostic Value of Respiratory System Compliance Under VV-ECMO on 180-day Mortality in COVID-19 ARDS.
Acronym: COMPLIECMO
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Matthieu KOSZUTSKI, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2022PI050
Record Dates: First submitted 2022-04-14; First posted 2022-04-22 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Ards; Mechanical Ventilation Pressure High; Extracorporeal Membrane Oxygenation
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No applicable — No applicable

SUMMARY:
Mortality of patients with COVID-19 associated acute respiratory distress syndrome (CARDS) treated with veno-venous extra-corporal membrane oxygenation (vv-ECMO) is increasing over time since the beginning of the COVID-19 pandemic. The objectives were to retrospectively describe over the first ten days after vv-ECMO implantation, the ventilatory management of CARDS and to assess the impact of static respiratory system compliance (CRS) on the first day of vv-ECMO on 180-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ARDS secondary to COVID-19 pneumonia requiring ECMO-VV support, hospitalized in the intensive care units of the CHRU of Nancy, Marseille or Bordeaux between 01/03/2020 and 31/12/2021.
* Age > 18 years old

Exclusion Criteria:

* Respiratory parameters not available on ten first day of VV ECMO implantation.
* Patient refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ARDS secondary to COVID-19 pneumonia requiring ECMO-VV support
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Vital status (dead or alive) | Days, 10.
  according to compliance during the first ten days of VV ECMO implantation

SECONDARY OUTCOMES:
Evolution of driving pressure | Days, 10
  after VV-ECMO implantation
Evolution of tidal volume | Days, 10
  after VV-ECMO implantation
Evolution of PEEP | days, 10
  after VV-ECMO implantation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No